CLINICAL TRIAL: NCT00548288
Title: Phase 1 Study of the Effect of Local Pamidronate Application in Preventing Periprosthetic Bone Loss After Total Cemented Hip Arthroplasty
Brief Title: Effect of Local Pamidronate in Preventing Bone Loss After Total Hip Arthroplasty
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: General and Teaching Hospital Celje (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAM19382CE
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Arthroplasty; Mineral Density
MeSH Terms: interventions — Pamidronate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: pamidronate

SUMMARY:
The aims of the study are to determine whether pamidronate applied locally causes diminished periprosthetic bone loss and decreased rate of bone turnover compared to patients receiving placebo after cemented total hip arthroplasty (THA). The study design will be prospective, randomized, and blind. Periprosthetic bone mineral density (BMD) will be measured with dual energy X-ray absorptiometry (DXA) at the total periprosthetic area as well as at seven Gruen zones or regions of interest. DXA scans will be performed at one week (baseline), three months, and six months postoperatively. Mean values of biochemical markers of bone turnover, BMD, and baseline-normalized BMD values will be compared between the bisphosphonate and placebo groups at each time point. For all temporal measurements including bone markers, BMD and normalized BMD, mean values will be compared across each time point within a given group.

ELIGIBILITY:
Inclusion Criteria:

* patients with hip arthritis scheduled for total cemented hip arthroplasty

Exclusion Criteria:

* pregnancy
* endoprosthesis on contralateral hip

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-11

PRIMARY OUTCOMES:
Periprosthetic bone mineral density | 6 months

SECONDARY OUTCOMES:
Biochemical markers of bone turnover | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Samo K Fokter, MD, PhD, Principal Investigator — General and Teaching Hospital Celje
Locations (1):
- Department for Orthopaedic Surgery and Sports Trauma, Celje Teaching Hospital, Celje, Slovenia